CLINICAL TRIAL: NCT06176521
Title: Evaluation of the Results of Laparoscopic Sacrohysteropexy and Sacrocolpopexy Surgeries Performed Without Mesh in the Surgical Treatment of Pelvic Organ Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GaziosmanpasaTREHs
Record Dates: First submitted 2023-12-09; First posted 2023-12-19 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2024-11

CONDITIONS: Pelvic Organ Prolapse
Keywords: sacrocolpopexy; sacrohysteropexy; pelvic organ prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Melanocyte-Stimulating Hormones

STUDY DESIGN:
Intervention Model Description: before and after surgery results of a single group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laparoscopic Sacrohysteropexy and Sacrocolpopexy Surgeries Performed Without Mesh (Other)
  Interventions: Procedure: Laparoscopic Sacrohysteropexy and Sacrocolpopexy Surgeries Performed Without Mesh

INTERVENTIONS:
Procedure: Laparoscopic Sacrohysteropexy and Sacrocolpopexy Surgeries Performed Without Mesh — Comparison of pre and postoperative POP-Q values of the patients undergone Laparoscopic Sacrohysteropexy and Sacrocolpopexy SurgeriesWithout Using Mesh Comparison of pre and postoperative PISQ-12 scores of the patients undergone Laparoscopic Sacrohysteropexy and Sacrocolpopexy Surgeries Without Using Mesh
  Other Names: Comparison of pre and postoperative POP-Q values of the patients undergone Laparoscopic Sacrohysteropexy and Sacrocolpopexy SurgeriesWithout Using Mesh; Comparison of pre and postoperative PISQ-12 scores of the patients undergone Laparoscopic Sacrohysteropexy and Sacrocolpopexy Surgeries Without Using Mesh

SUMMARY:
Evaluation of the anatomical and functional results of laparoscopic sacrohysteropexy and sacrocolpopexy surgeries performed without using mesh in the surgical treatment of pelvic organ prolapse

ELIGIBILITY:
Inclusion Criteria:

1. being 18 years old or older
2. needing an operation for symptomatic pelvic organ prolapse -

Exclusion Criteria:

1. past history of chemotherapy or radiotherapy
2. past history of pelvic organ prolapse surgery
3. if there is a contraindication of laparoscopy -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Pre and post operative assessment of POP-Q measurements | 1 year
  POP-Q values of patients before and after laparoscopic Sacrohysteropexy and Sacrocolpopexy Surgeries Performed Without Mesh on Pelvic Organ Prolapse will be compared.
Pre and post operative assessment of Pelvic Organ Prolapse / Incontinence Sexual | 1 year
  Units on a scale of the patients obtained with Pelvic Organ Prolapse / Incontinence Sexual Questionnaire (PISQ-12) will be compared before and after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpasa Training and Research Hospital, Istanbul, Turkey (Türkiye)